CLINICAL TRIAL: NCT04063592
Title: A Novel Approach to Lower Extremity Residual Limb Revision to Augment Volitional Motor Control, Restore Proprioception and Reverse Limb Atrophy
Brief Title: AMI Construction in Lower Extremity Residual Limbs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Massachusetts Institute of Technology (Other); Walter Reed National Military Medical Center (U.S. Federal Agency); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Matthew Carty, Principal Investigator, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019P001681; CDMRP-180114 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2019-06-15; First posted 2019-08-21 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Amputation
Keywords: Amputation; Residual limb pain; Phantom pain; Residual limb atrophy; Prosthesis control
MeSH Terms: conditions — Phantom Limb

STUDY DESIGN:
Intervention Model Description: Prospective clinical trial in which intervention subjects will serve as their own control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Subjects undergoing the proposed operative intervention. Intervention patients will serve as their own control for all outcome measures
  Interventions: Procedure: Residual limb revision

INTERVENTIONS:
Procedure: Residual limb revision — Surgical procedure involving construction of agonist-antagonist myoneural interfaces (AMIs)

SUMMARY:
This study will involve the development of a novel approach to lower extremity residual limb surgical revision that offers the promise of augmenting volitional motor control, restore proprioception and reverse atrophy

DETAILED DESCRIPTION:
The hypothesis of this research protocol is that we will be able to modify the residual limbs of patients who have already undergone lower extremity amputations so as to include biological actuators that will enable the successful employment of next generation lower extremity prostheses, diminish/eliminate phantom limb pain, restore proprioception and regenerate lost muscle mass. The specific aims of the project are as follows:

1. To develop a standardized operative technique for both above knee (AK) and below knee (BK) amputation revision procedures that includes AMIs to restore musculotendinous proprioceptive capabilities
2. To assess the capacity for these actuators to provide enhanced motor control and sensory feedback, as well as ablate phantom limb symptomatology and augment residual limb muscle mass
3. To determine the reinnervation time course and longevity of these biological constructs
4. To validate the functional and somatosensory superiority of the proposed revision technique over standard approaches to BKA and AKA
5. To develop a modified acute postoperative rehabilitation strategy suited to this new surgical approach

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-65
* Has already undergone a standard AKA or BKA procedure
* Suffers from symptoms such as:

  * Intractable pain
  * Deterioration of skin on or around stump
  * Suffering from other sources of discomfort arising from stump
* Intact inherent wound healing
* Adequate communication skills
* High motivation

Exclusion Criteria:

* Inadequate health to undergo operative procedure using standard anesthesia (i.e. cardiopulmonary)
* Individuals with impaired wound healing
* Individuals suffering from extensive peripheral neuropathies
* Active smokers
* Individuals with a history of poor compliance
* Women who are pregnant or plan to become pregnant before surgical intervention

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2020-02-24 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Limb Morphology and Changes in Muscle Volume | Years 1-3
  Clinical examination and images from CT/MRI will be combined to construct a holistic view of the morphology of the residual limb. Imaging studies and limb measurements taken in clinic will also be used to measure muscle atrophy/hypertrophy over time.
Degree of Motor Activation of AMI Muscles and Volitional Control of Phantom Limb | Years 1-3
  Clinical examination will confirm the sliding motion of the AMI constructs with radiologic evaluation measuring the length of muscle excursion through each construct. Functional testing and testing using a prosthesis will determine how well a patient is able to volitionally control the AMI muscles.
Evidence of Proprioception | Years 1-3
  Subjective reporting combined with tests run using a prosthesis will indicate if proprioception is still intact after surgery. Results will be confirmed by monitoring brain activity during limb movement activities via fMRI.
Evidence of Sensory Perception | Years 1-3
  Subjective reporting and clinical tests of Semmes-Weinstein and two-point discrimination will determine if the patient has sensory perception on the residual limb.
General Health | Years 1-3
  Patient-reported outcomes metrics from five validated tests (SIP136, EQ-5D, SF-36, LEFS, PROMIS) will be combined to create an overall picture of patients' general health during and after their recovery.
Complications | Years 1-3
  Delayed wound healing, infection, need for additional surgery, PE/DVT, death

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Carty, MD, Principal Investigator — Brigham and Women's Hospital
Locations (3):
- United States (3):
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Massachusetts Institute of Technology, Cambridge, Massachusetts

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be available to other researchers